CLINICAL TRIAL: NCT03069716
Title: A Mobile Health Intervention in Pulmonary Arterial Hypertension
Acronym: mHealth
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Vanderbilt University Medical Center (Other)
Collaborators: Johns Hopkins University (Other)
Responsible Party: Principal Investigator, Evan Brittain, Assistant Professor of Medicine, Vanderbilt University Medical Center
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: IRB #162004
Record Dates: First submitted 2017-02-21; First posted 2017-03-03 (Actual); Results first posted 2021-06-24 (Actual); Last update posted 2021-06-25 (Actual); Status verified 2021-06

CONDITIONS: Pulmonary Arterial Hypertension; Idiopathic Pulmonary Arterial Hypertension; Heritable Pulmonary Arterial Hypertension; Associated Pulmonary Arterial Hypertension
Keywords: Pulmonary Arterial Hypertension
MeSH Terms: conditions — Pulmonary Arterial Hypertension; Familial Primary Pulmonary Hypertension

STUDY DESIGN:
Intervention Model Description: Randomization will occur after a two-week run-in period to improve ability to identify a true baseline step count and account for potential dropout. Participants will be assigned to either the smartphone text messaging or no smartphone text messaging arms in a random manner until 25 participants are enrolled into each arm. Permuted block randomization stratified by functional class (I/II vs. III) will be used to ensure approximate balance of treatment groups within each stratum over time. Randomization will be performed in small blocks, which vary in size. Investigators will be unaware of the size or order of the blocks. Randomization will occur through REDCap by a study coordinator. Although the texting intervention will end after Week 12, subjects in both groups will be asked to continue wearing the Fitbit Charge HR device for an additional 3 weeks to determine whether withdrawal of the texting intervention results in a reduction in step counts.
Who Masked: Care Provider, Investigator, Outcomes Assessor
Masking Description: Investigators are blinded.
  Study personnel conducting 6MWT and echo will be blinded.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Smartphone Text Messaging (Experimental): Group receives personalized, health coaching via "smart" text messages.
  Interventions: Device: Smartphone Text Messaging; Device: Fitbit Charge HR
- No Smartphone Text Messaging (Other): Group does not receive personalized, health coaching via "smart" text messages.
  Interventions: Device: Fitbit Charge HR

INTERVENTIONS:
Device: Smartphone Text Messaging — A HIPPA compliant text messaging platform is linked to the Fitbit Application Program Interface. Real time activity data will be transmitted from the subject's smartphone to our mHealth platform via cellular network. Subjects will receive 3 texts/day in sync with their preferred morning, lunch, and evening leisure schedule (defined at enrollment). These texts will use personal, disease-specific, and provider information to deliver 2 types of messages customized to the current step count and sent in equal proportion. Messages are designed to facilitate self-awareness, reinforce step targets, and link physical activity with a reward or memorable cue.
  Other Names: mHealth activity intervention
  Arms: Smartphone Text Messaging
Device: Fitbit Charge HR — The Fitbit Charge HR tri-axial accelerometer will be used to continuously gather data on physical activity, heart rate, and sleep. This device provides feedback in units of activity (steps, stairs climbed, activity time, and exercise time) and heart rate (per second when active, per 5 seconds when inactive). It has been validated against research devices in free-living conditions and is relatively inexpensive.
  Other Names: Digital Activity Tracker

SUMMARY:
This study proposes the use of a mobile health intervention (utilizing a smart phone app) to encourage increased exercise in PAH patients. The study will be a randomized trial to examine feasibility of an mHealth (mobile device) Fitbit Charge HR and cell phone application intervention to improve step counts and increase participants activity level as compared to no intervention. The Fitbit Charge Heart Rate (HR) monitors activity and the cell phone application provides encouragement notifications to half the subjects while the other half do not receive encouragements.

DETAILED DESCRIPTION:
Patients with pulmonary arterial hypertension (PAH) have severely reduced exercise capacity and reduced quality of life. At diagnosis, most PAH patients are New York Heart Association (NYHA) functional class III with symptoms of fatigue and shortness of breath with less than ordinary activity. Physical activity confers multiple benefits relevant to PAH pathophysiology including improvements in endothelial function, energy metabolism, and right ventricular (RV) function. Increasing physical activity is highly efficacious in PAH, resulting in six-minute walk distance (6MWD) improvement that exceeds the effect of medications.

The goal of this proposal is to adapt and test the feasibility of our mHealth intervention to increase physical activity in a geographically diverse PAH population. In secondary aims, we will assess conventional PAH trial outcomes (6MWD, quality of life) and physiologic mechanisms by which increasing activity may improve exercise capacity.

The investigator hypothesizes that an mHealth intervention is feasible and will increase physical activity in subjects with PAH. This study proposes a randomized trial of unblinded step tracking with smart texts tracking for 12 weeks. Participants will wear a display-free triaxial accelerometer, which will continuously transmit data to a compatible smartphone (owned by 75% of our PAH population). Efficacy endpoints have been selected to mirror FDA criteria for drug approval in PAH. The following aims will be tested:

Aim 1: To test the feasibility of an mHealth intervention to increase step counts in patients with PAH. Fifty PAH patients will be randomized to the mHealth intervention or usual activity for 12 weeks. The primary endpoint will be daily step count during Week 12. Secondary endpoints will assess step target achievement, daily activity time, and aerobic time. The fidelity of data collection and text transmission will also be assessed.

Aim 2: To examine the effect of an mHealth intervention on exercise capacity and quality of life. Participants will complete a six minute walk test and the emPHasis-10 questionnaire at baseline and 12 weeks. The primary endpoint will be six minute walk distance. Secondary endpoints will be emPHasis-10 quality of life scale score, Borg dyspnea score, and resting heart rate.

Aim 3: To examine the effect of an mHealth intervention on mechanisms of improved exercise capacity. Subjects will undergo echocardiography, blood draw, and body composition assessment. The primary endpoint will be RV longitudinal strain. Secondary endpoints will be the homeostatic model assessment of insulin resistance, lean muscle and fat mass, and B-type natriuretic peptide.

ELIGIBILITY:
Inclusion Criteria:

1. Aged 18 or older.
2. Diagnosed with idiopathic, heritable, or associated (connective tissue disease, drugs, or toxins) pulmonary arterial hypertension (PAH) according to World Health Organization consensus recommendations.
3. Stable PAH-specific medication regimen for three months prior to enrollment. Subjects with only a single diuretic adjustment in the prior three months will be included.
4. Subjects must own a Bluetooth capable modern smartphone capable of receiving and sending text messages and an active data plan.

Exclusion Criteria:

1. Prohibited from normal activity due to wheelchair bound status, bed bound status, reliance on a cane/walker, activity-limiting angina, activity-limiting osteoarthritis, or other condition.
2. Pregnancy.
3. Diagnosis of PAH etiology other than idiopathic, heritable, or associated.
4. Forced vital capacity <70% predicted.
5. Functional class IV heart failure.
6. Requirement of > 1 diuretic adjustment in the prior three months.
7. Preferred form of activity is not measured by an activity tracker (swimming, yoga, ice skating, stair master, or activities on wheels such as bicycling or rollerblading).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 49 (Actual)
Dates: Start 2017-08-02 (Actual); Primary Completion 2020-04-24 (Actual); Study Completion 2020-04-24 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Evan Brittain, MD, MSc, Principal Investigator — Vanderbilt University Medical Center
Locations (1):
- Vanderbilt University Medical Center, Nashville, Tennessee, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Martin SS, Feldman DI, Blumenthal RS, Jones SR, Post WS, McKibben RA, Michos ED, Ndumele CE, Ratchford EV, Coresh J, Blaha MJ. mActive: A Randomized Clinical Trial of an Automated mHealth Intervention for Physical Activity Promotion. J Am Heart Assoc. 2015 Nov 9;4(11):e002239. doi: 10.1161/JAHA.115.002239. PMID 26553211
- [Background] Pugh ME, Buchowski MS, Robbins IM, Newman JH, Hemnes AR. Physical activity limitation as measured by accelerometry in pulmonary arterial hypertension. Chest. 2012 Dec;142(6):1391-1398. doi: 10.1378/chest.12-0150. PMID 22576635
- [Background] Bravata DM, Smith-Spangler C, Sundaram V, Gienger AL, Lin N, Lewis R, Stave CD, Olkin I, Sirard JR. Using pedometers to increase physical activity and improve health: a systematic review. JAMA. 2007 Nov 21;298(19):2296-304. doi: 10.1001/jama.298.19.2296. PMID 18029834
- [Background] Mereles D, Ehlken N, Kreuscher S, Ghofrani S, Hoeper MM, Halank M, Meyer FJ, Karger G, Buss J, Juenger J, Holzapfel N, Opitz C, Winkler J, Herth FF, Wilkens H, Katus HA, Olschewski H, Grunig E. Exercise and respiratory training improve exercise capacity and quality of life in patients with severe chronic pulmonary hypertension. Circulation. 2006 Oct 3;114(14):1482-9. doi: 10.1161/CIRCULATIONAHA.106.618397. Epub 2006 Sep 18. PMID 16982941
- [Derived] Hemnes AR, Silverman-Lloyd LG, Huang S, MacKinnon G, Annis J, Whitmore CS, Mallugari R, Oggs RN, Hekmat R, Shan R, Huynh PP, Yu C, Martin SS, Blaha MJ, Brittain EL. A Mobile Health Intervention to Increase Physical Activity in Pulmonary Arterial Hypertension. Chest. 2021 Sep;160(3):1042-1052. doi: 10.1016/j.chest.2021.04.012. Epub 2021 Apr 17. PMID 33878341

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: After participant is enrolled, they are given a fitbit device to wear for a 14 day run-in period leading up to the baseline visit. After the baseline visit is completed they are then randomized.
  Reasons why a participants may have been removed from study prior to randomization include the participant dropping out for personal or medical issues.
Groups:
- Run-in Participants: participant is enrolled, they are given a fitbit device to wear for a 14 day run-in period leading up to the baseline visit.
Period: Run-in Period (2 Weeks)
Arm/Group | Run-in Participants | Smartphone Text Messaging | No Smartphone Text Messaging
Started | 49 | 0 | 0
Completed | 42 | 0 | 0
Not Completed | 7 | 0 | 0
Not completed — Adverse Event | 1 | 0 | 0
Not completed — Protocol Violation | 1 | 0 | 0
Not completed — Withdrawal by Subject | 5 | 0 | 0
Period: Randomized Treatment
Arm/Group | Run-in Participants | Smartphone Text Messaging | No Smartphone Text Messaging
Started | 0 | 20 | 22
Completed | 0 | 18 | 22
Not Completed | 0 | 2 | 0
Not completed — Withdrawal by Subject | 0 | 2 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Smartphone Text Messaging | No Smartphone Text Messaging | Total
Number analyzed (Participants) | 20 | 22 | 42
Age, Continuous [Median (Inter-Quartile Range); unit: Years] | 47 [41 to 54] | 47 [36 to 58] | 47 [39 to 57]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15 | 21 | 36
  Male | 5 | 1 | 6
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 1
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 6 | 3 | 9
  White | 13 | 19 | 32
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Daily Step Count
Description: Change from baseline mean daily step count at week 12.
Time Frame: Baseline to 12 weeks
Measure: Median (Inter-Quartile Range); unit: Steps
Arm/Group | Smartphone Text Messaging | No Smartphone Text Messaging
Number analyzed (Participants) | 18 | 22
Steps | 1409 [-32 to 2220] | -149 [-1010 to 735]

2. Secondary Outcome: Six Minute Walk Test Distance
Description: Change from baseline of six minute walk test distance (meters) at week 12.
Time Frame: Baseline to 12 weeks
Population: Only 17 participants in the Smartphone Text Messaging arm were analyzed due to research shut downs during COVID. Any assessments requiring an in-person visit were not completed for one participant.
Measure: Median (Inter-Quartile Range); unit: meters
Arm/Group | Smartphone Text Messaging | No Smartphone Text Messaging
Number analyzed (Participants) | 17 | 22
meters | 3 [-42 to 23] | -6 [-36 to 26]

3. Secondary Outcome: Right Ventricle (RV) Strain
Description: Change from baseline of RV free wall longitudinal strain at week 12.
Time Frame: Baseline to 12 weeks
Population: as for outcome 2
Measure: Median (Inter-Quartile Range); unit: percentage of deformation
Arm/Group | Smartphone Text Messaging | No Smartphone Text Messaging
Number analyzed (Participants) | 17 | 22
percentage of deformation | -0.1 [-1.6 to 2.0] | 0.4 [-1.9 to 1.8]

4. Secondary Outcome: Percentage of Days Participants Met Their Daily Step Count Goal
Description: All participants were provided with an Fitbit Charge Heart Rate mobile device to monitor daily step counts, activity time, and aerobic time. The daily goal was communicated via text to the intervention group and was the baseline step count average for the control group. Increased daily goal attainment indicates increased activity level
Time Frame: Baseline to 12 weeks
Measure: Number; unit: percent of days at goal across group
Arm/Group | Smartphone Text Messaging | No Smartphone Text Messaging
Number analyzed (Participants) | 18 | 22
percent of days at goal across group | 41 | 24

5. Secondary Outcome: Daily Aerobic Time
Description: Change in minutes of activity per day between Week 12 and Baseline
Time Frame: Baseline to 12 weeks
Measure: Median (Inter-Quartile Range); unit: minutes
Arm/Group | Smartphone Text Messaging | No Smartphone Text Messaging
Number analyzed (Participants) | 18 | 22
minutes | 10 [-36 to 58] | -16 [-44 to 29]

6. Secondary Outcome: Change From Baseline at Week 12 in emPHasis-10 Questionnaire Score
Description: Quality of life was assessed using the emPHasis-10 questionnaire, a disease-specific self-administered 10-question questionnaire designed for routine assessment of health-related quality of life in pulmonary hypertension. Total score can range from 0 to 50, with higher scores indicating a worse quality of life. Change from Baseline was calculated as the value at Week 12 minus the value at Baseline. The Week 12 value was defined as the last assessment at or prior to Week 12.
Time Frame: Baseline to 12 weeks
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | Smartphone Text Messaging | No Smartphone Text Messaging
Number analyzed (Participants) | 18 | 22
units on a scale | -3 [-4.8 to 3.0] | 1.0 [-2.0 to 3.5]

7. Secondary Outcome: Change From Baseline on the SF-36 Mental Component Summary (MCS) Score
Description: SF-36 consists of 36 questions measuring 8 health domains: physical functioning, bodily pain, role limitations due to physical problems, role limitations due to emotional problems, general health perceptions, mental health, social function, and vitality. The patient's responses are solicited using Likert scales that vary in length, with 3-6 response options per item. The SF-36 can be scored into the 8 health domains named above and two overall summary scores: physical component summary (PCS) and mental component summary (MCS) scores. The domain and summary scores range from 0 to 100; higher scores indicate better levels of function and/or better health
Time Frame: Baseline to 12 weeks
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | Smartphone Text Messaging | No Smartphone Text Messaging
Number analyzed (Participants) | 18 | 22
units on a scale | 3.8 [0.9 to 8.7] | 1.5 [-9.3 to 3.3]

8. Secondary Outcome: Change From Baseline to Week 12 in Borg Dyspnea Score
Description: The Borg Dyspnea score is a self-rating scale to evaluate the severity of dyspnea (from 0 "no shortness of breath at all" to 10 "very, very severe / maximal" shortness of breath). The scale was completed at the beginning and conclusion of each 6-minute walk test at baseline and at Week 12. Median change from baseline in scoring was reported.
Time Frame: Baseline to 12 weeks
Population: as for outcome 2
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | Smartphone Text Messaging | No Smartphone Text Messaging
Number analyzed (Participants) | 17 | 22
units on a scale | -1.0 [-2.0 to 0.0] | 0.0 [-1.0 to 0.0]

9. Secondary Outcome: Resting Heart Rate
Description: Change in heart rate between Week 12 and Baseline
Time Frame: Baseline to 12 weeks
Measure: Median (Inter-Quartile Range); unit: beats per minute
Arm/Group | Smartphone Text Messaging | No Smartphone Text Messaging
Number analyzed (Participants) | 18 | 22
beats per minute | 0 [-7 to 4] | 0 [-7 to 7]

10. Secondary Outcome: Total Lean Mass
Description: Change from baseline lean mass at week 12.
Time Frame: Baseline to 12 weeks
Population: as for outcome 2
Measure: Median (Inter-Quartile Range); unit: kilograms
Arm/Group | Smartphone Text Messaging | No Smartphone Text Messaging
Number analyzed (Participants) | 17 | 22
kilograms | 0.1 [-1.1 to 1.2] | 0.0 [-0.6 to 1.1]

11. Secondary Outcome: Insulin Resistance
Description: Insulin resistance measured by the Homeostatic Model Assessment for Insulin Resistance insulin resistance score (HOMA-IR) utilizing the formula: fasting plasma glucose (mmol/l) times fasting serum insulin (mU/l) divided by 22.5. Low HOMA-IR values indicate high insulin sensitivity, whereas high HOMA-IR values indicate low insulin sensitivity (insulin resistance).
Time Frame: Baseline to 12 weeks
Population: as for outcome 2
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | Smartphone Text Messaging | No Smartphone Text Messaging
Number analyzed (Participants) | 17 | 22
units on a scale | 0.3 [-0.2 to 0.8] | 0.0 [-0.6 to 0.1]

12. Secondary Outcome: BNP
Description: Change from baseline B-type natriuretic peptide level at week 12.
Time Frame: Baseline to 12 weeks
Population: as for outcome 2
Measure: Median (Inter-Quartile Range); unit: pg/mL
Arm/Group | Smartphone Text Messaging | No Smartphone Text Messaging
Number analyzed (Participants) | 17 | 22
pg/mL | -2 [-13 to 1] | 7 [-14 to 22]

13. Secondary Outcome: Change From Baseline on the SF-36 Physical Component Summary (PCS) Score
Description: as for outcome 7
Time Frame: Baseline to 12 weeks
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | Smartphone Text Messaging | No Smartphone Text Messaging
Number analyzed (Participants) | 18 | 22
units on a scale | -0.8 [-3.6 to 1.5] | -0.4 [-3.3 to 3.5]

14. Secondary Outcome: Minutes of Moderate-vigorous Activity
Description: Change in minutes between Week 12 and Baseline
Time Frame: Baseline to 12 Weeks
Measure: Median (Inter-Quartile Range); unit: minutes
Arm/Group | Smartphone Text Messaging | No Smartphone Text Messaging
Number analyzed (Participants) | 18 | 22
minutes | 1.6 [-5.1 to 16.1] | -0.6 [-4.5 to 1.4]

15. Secondary Outcome: Visceral Fat Volume
Description: Change in fat volume between Week 12 and Baseline
Time Frame: Baseline to Week 12
Population: as for outcome 2
Measure: Median (Inter-Quartile Range); unit: mL
Arm/Group | Smartphone Text Messaging | No Smartphone Text Messaging
Number analyzed (Participants) | 17 | 22
mL | -67 [-432 to 0.0] | 21 [-84 to 177]

ADVERSE EVENTS:
Time Frame: Adverse Event data collected for 12 weeks from each participant
Description: Definitions of an adverse event and/or serious adverse event, used to collect adverse event information, is in line with clinicaltrials.gov.
Arm/Group | Smartphone Text Messaging | No Smartphone Text Messaging
All-Cause Mortality (participants affected / at risk) | 0/20 | 0/22
Serious Adverse Events (participants affected / at risk) | 2/20 | 0/22
Other Adverse Events (participants affected / at risk) | 5/20 | 4/22
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Smartphone Text Messaging (N=20) | No Smartphone Text Messaging (N=22)
Hypertensive urgency (Cardiac disorders) | 1 (1) | 0 (0)
Medication escalation (Respiratory, thoracic and mediastinal disorders) | 1 (1) | NA
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Smartphone Text Messaging (N=20) | No Smartphone Text Messaging (N=22)
Chest Pain (Cardiac disorders) | 4 (7) | 1 (1)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 3 (4)
Edema (Cardiac disorders) | 2 (5) | 4 (12)
Fatigue (General disorders) | 2 (3) | 4 (7)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-08-06): https://cdn.clinicaltrials.gov/large-docs/16/NCT03069716/Prot_SAP_000.pdf